CLINICAL TRIAL: NCT05754736
Title: Efficacy and Safety of Ametinib Combined With Bevacizumab in First-line Treatment of Non-oligometastatic Advanced NSCLC With EGFR-mutations.
Brief Title: Clinical Study of Ametinib Combined With Bevacizumab in First-line Treatment of Advanced NSCLC With EGFR-mutations.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-005
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ametinib combined with bevacizumab (Experimental): Ametinib 110 mg po qd bevacizumab 15mg/kg ivdrip q3w
  Interventions: Drug: Ametinib combined with bevacizumab

INTERVENTIONS:
Drug: Ametinib combined with bevacizumab — Ametinib 110mg po qd bevacizumab 15mg/kg ivdrip q3w
  Other Names: Third-generation TKI combined with antivascular targeting drug

SUMMARY:
To explore the intracranial/extracranial ORR, PFS, QoL, safety, dynamic changes of tissue, cerebrospinal fluid, and plasma DNA in patients with newly diagnosed advanced NSCLC with EGFR mutation with/without brain metastasis given first-line treatment with almonertinib combined with bevacizumab at the initial stage of treatment, during treatment and after drug resistance, and the correlation between early clearance of sensitive mutations and survival.

DETAILED DESCRIPTION:
This is a one-arm prospective study to evaluate the first-line treatment of amitinib in combination with bevacizumab in patients with advanced NSCLC with EGFR mutations Effectiveness and safety. Subjects received amitinib and bevacizumab during the treatment cycle and were evaluated for efficacy every 6-8 weeks. Subject receives medication until disease progression, intolerable toxicity, or withdrawal of informed consent. The primary endpoint was progression-free survival as measured by the solid tumor Response Assessment Criteria (RECIST v1.1). Primary endpoints included objective response rate (ORR), progression-free period (PFS), and secondary endpoints included objective response rate (iORR), progression-free period (iPFS), overall survival (OS), quality of life (QoL), and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years old and ≤75years old;

  * Non-squamous non-small cell lung cancer (NSCLC) confirmed by pathology (including histology or cytology); ③ EGFR mutation positive (exon 19 deletion or exon 21 L858R mutation); (4) ≥3 intracranial metastases, asymptomatic brain metastases; (5) Never received antitumor therapy before;

    * There was at least 1 measurable intracranial and extracranial lesion in CT/MRI according to RECIST1.1 criteria.

      ⑦ Predicted survival ≥3 months;

      ⑧ ECOG score 0-1;

      ⑨ The main organs (liver, kidney, heart) function normally.

      ⑩ Sign informed consent forms.

Exclusion Criteria:

* The intracranial metastases were oligometastases;

  * There are symptoms of increased intracranial pressure; (3) Previous or co-existing malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix); (4) Patients with hypertension and can not be reduced to the normal range after antihypertensive drug treatment, have grade I coronary heart disease, grade I arrhythmia and grade I cardiac insufficiency;

    * Patients with definite tendency to gastrointestinal bleeding; ⑥ with hemoptysis symptoms; ⑦ Abnormal coagulation function (INR>1.5, APTT>1.5 ULN), with bleeding tendency; ⑧ Have a history of psychotropic drug abuse and can not abstain or have mental disorders; ⑨According to the investigator's judgment, Patients who have a serious concomitant disease that endangers the patient's safety or affects the patient's completion of the study, and who have previous or current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severe impairment of lung function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  It refers to the proportion of patients (mainly solid tumors) whose tumor has shrunk to a certain extent and remained there for a certain period of time, including Complete Response (CR) and Partial Response (PR)
Progression Free Survival | 2 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Intracranial Objective Response Rate | 2 year
  It refers to the proportion of patients with brain metastases，whose Intracranial tumor has shrunk to a certain extent and remained there for a certain period of time, including Complete Response (CR) and Partial Response (PR)
Intracranial Progression Free Survival | 2 year
  The length of time during and after the treatment of lung cancer, that a patient with brain metastases lives with the tumor but it does not get worse
Overall Survival | 3 year
  Time from randomization to death from any cause
Quality of life score | 3 year
  Quantitative scoring system for patients' self-subjective self-assessment of current symptom tolerance
Adverse event | 3 year
  It refers to all adverse medical events that occur after a subject receives an investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug
  It refers to all adverse medical events that occur after a subject receives an investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug
  It refers to all adverse medical events that occur after a subject receives an investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University
Locations (1):
- The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramotar M, Barnes S, Moraes F, Dasgupta A, Laperriere N, Millar BA, Berlin A, Conrad T, van Prooijen M, Damyanovich A, Heaton R, Cho YB, Coolens C, Liu G, Shepherd FA, Bradbury P, Leighl N, Bernstein M, Zadeh G, Kongkham P, Doherty M, Shultz DB. Neurological Death is Common in Patients With EGFR Mutant Non-Small Cell Lung Cancer Diagnosed With Brain Metastases. Adv Radiat Oncol. 2019 Nov 26;5(3):350-357. doi: 10.1016/j.adro.2019.11.002. eCollection 2020 May-Jun. PMID 32529128
- [Result] Yoneda K, Imanishi N, Ichiki Y, Tanaka F. Treatment of Non-small Cell Lung Cancer with EGFR-mutations. J UOEH. 2019;41(2):153-163. doi: 10.7888/juoeh.41.153. PMID 31292359
- [Result] Passiglia F, Pilotto S, Facchinetti F, Bertolaccini L, Del Re M, Ferrara R, Franchina T, Malapelle U, Menis J, Passaro A, Ramella S, Rossi G, Trisolini R, Novello S. Treatment of advanced non-small-cell lung cancer: The 2019 AIOM (Italian Association of Medical Oncology) clinical practice guidelines. Crit Rev Oncol Hematol. 2020 Feb;146:102858. doi: 10.1016/j.critrevonc.2019.102858. Epub 2019 Dec 28. PMID 31918343